CLINICAL TRIAL: NCT06965881
Title: A Phase 1, Open-label, 2-part Study to Evaluate the Pharmacokinetics and Safety Effects Following Coadministration of a CYP3A4 Inducer (Carbamazepine) or Inhibitor (Itraconazole), With Radiprodil in Healthy Adult Participants
Brief Title: Study to Evaluate the Pharmacokinetics and Safety Effects Following Coadministration of Carbamazepine or Itraconazole With Radiprodil in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to the lack of operational capabilities of the sites to segregate participants as needed.
Sponsor: GRIN Therapeutics, Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-GRIN-504
Record Dates: First submitted 2025-04-11; First posted 2025-05-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Tuberous Sclerosis Complex (TSC); Focal Cortical Dysplasia; Other Neurological Disorders
Keywords: healthy adults; tuberous sclerosis; focal cortical dysplasia
MeSH Terms: conditions — Tuberous Sclerosis; Focal Cortical Dysplasia | interventions — radiprodil; Carbamazepine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Radiprodil with Carbamazepine (Experimental): Participants will receive multiple oral doses of Radiprodil with Carbamazepine to evaluate the effect that carbamazepine may have on Radiprodil.
  Interventions: Drug: Radiprodil with Carbamazepine
- Part B: Radiprodil with Itraconazole (Experimental): Participants will receive multiple oral doses of Radiprodil with Itraconazole to evaluate the effect that itraconazole may have on Radiprodil.
  Interventions: Drug: Radiprodil with Itraconazole

INTERVENTIONS:
Drug: Radiprodil with Carbamazepine — Participants will receive oral doses of Radiprodil in the range of 7.5mg to 30mg along with oral doses of Carbamazepine in the range of 100mg to 300mg twice daily over a period of 27 days.
  Arms: Part A: Radiprodil with Carbamazepine
Drug: Radiprodil with Itraconazole — Participants will receive oral doses of Radiprodil in the range of 7.5mg to 15mg along with oral doses of Itraconazole 200mg twice daily over a period of 21 days.
  Arms: Part B: Radiprodil with Itraconazole

SUMMARY:
This is a Phase 1, open-label, 2-part study to evaluate the effect of multiple doses of oral carbamazepine or oral itraconazole on the plasma pharmacokinetic profile of radiprodil in healthy adult participants. In addition, the safety and tolerability of radiprodil given together with oral carbamazepine or itraconazole will be assessed.

DETAILED DESCRIPTION:
This is an open label study conducted in healthy adult volunteers. The study will be conducted in 2 parallel parts. A total of 36 participants will be enrolled in the study (N=18 per Part).

Part A: will enrol 18 participants to receive multiple oral doses of the radiprodil in the range of 7.5mg to 30mg with oral carbamazepine.

Part B: will enrol 18 participants to receive multiple oral doses of radiprodil in the range of 7.5mg to 15mg with oral itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18 and 55 years of age, inclusive, at Screening
* Body mass index (BMI) between 18 and 32 kg/m2 (inclusive) and weighs at least 50 kg at Screening
* Medically healthy in the opinion of the PI or delegate
* Female participants must be non-lactating and of non-child-bearing potential; or if child-bearing potential must agree to not to attempt to become pregnant or donate ova from signing consent until at least 90 days after the last dose of study drug and must agree to use adequate contraception
* Male participants must agree to not donate sperm from signing consent until at least 90 days after the last dose of study drug and must agree to use adequate contraception
* Have suitable venous access for blood sampling.
* Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions

Exclusion Criteria:

* Known hypersensitivity to the study drug or any of the study drug ingredients
* Genetic testing positive for HLA genotypes
* Has a history of severe allergic or anaphylactic reaction
* Has history of surgery in the past 90 days prior to Day 1
* Has a history of of risk factors for torsade de pointes or a known arrythmia
* Has a history of or positive serology for HIV, Hepatitis B or Hepatitis C virus at Screening.
* Has a history of suicide attempts or deliberate self-harm
* Use of cannabidiol (CBD) within 30days of Day -1
* Regular consumption of more than 10 standard alcoholic drinks/week and/or more than 4 standard alcoholic drinks on any one day
* Routine consumption of an average of more than five (5) 240 mL servings of coffee or other caffeinated beverages per day
* Use of tobacco-containing products and nicotine or nicotine containing products in the 2 months prior to Day -1
* Women of childbearing potential using oral, injected or implanted hormonal contraception
* Has any other condition or prior therapy that, in the opinion of the Investigator or delegate, may potentially compromise the safety or compliance of the participant, or may preclude the participant from successfully completing the study.

Other inclusion/exclusion eligibility criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Part A: To assess the effect of oral carbamazepine on the maximum observed plasma concentration (Cmax) of oral dosing of radiprodil | Blood samples will be collected on Days 7 to 10 and 25 to 28.
Part B: To assess the effect of oral itraconazole on the maximum plasma concentration (Cmax) of oral dosing of radiprodil | Blood samples will be collected Days 5 to 9 and 18 to 22.
Part A: To asses the effect of oral carbamazepine on radiprodil area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) | Blood samples will be collected on Days 7 to 10 and 25 to 28.
Part B: To asses the effect of oral itraconazole on the radiprodil area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) | Blood samples will be collected Days 5 to 9 and 18 to 22.
Part A: To assess the effect of oral oral carbamazepine on the area under the plasma concentration-time curve to the end of dosing interval (AUCtau) of oral dosing of radiprodil | Blood samples will be collected on Days 7 to 10 and 25 to 28
Part B: To assess the effect of oral itraconazole on the area under the plasma concentration-time curve to the end of dosing interval (AUCtau) of oral dosing of radiprodil | Blood samples will be collected Days 5 to 9 and 18 to 22

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs), TEAEs Leading to Discontinuation and Severity of TEAEs | From Screening to Day 30 and follow up visit 30 days post last dose
  Frequency, type, severity and duration of adverse events, serious adverse events and adverse drug reactions.
Part A: To assess the area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) of carbamazepine and carbamazepine metabolites following oral dosing of carbamazepine alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 18 and 25.
Part B: To assess the area under the plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) of itraconazole following oral dosing of itraconazole alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 13 and 18.
Part B: To assess the area under the plasma concentration-time curve to the end of dosing interval (AUCtau) of itraconazole following oral dosing of itraconazole alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 13 and 18.
Part A: To assess the area under the plasma concentration-time curve to the end of dosing interval (AUCtau) of carbamazepine and carbamazepine metabolites following oral dosing of carbamazepine alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 18 and 25.
Part A: To assess the time to maximum observed plasma concentration (Tmax) of carbamazepine and carbamazepine metabolites following oral dosing of carbamazepine alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 18 and 25.
Part B: To assess the time to maximum observed plasma concentration (Tmax) of itraconazole following oral dosing of itraconazole alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 13 and 18.
Part B: To assess the maximum observed plasma concentration (Cmax) of itraconazole following oral dosing of itraconazole alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 13 and 18.
Part A: To assess the maximum observed plasma concentration (Cmax) of carbamazepine and carbamazepine metabolites following oral dosing of carbamazepine alone and in the presence of radiprodil | Blood samples for plasma PK will be collected on Days 18 and 25.
Number of participants with abnormal laboratory test results | From Screening to Day 30 and follow up visit 30 days post last dose
  The clinical laboratory tests include hematology, serum chemisty and coagulation
To assess the Columbia-Suicide Severity Rating Scale (C-SSRS) scores | From Screening to Day 30 and follow up visit 30 days post last dose
  The C-SSRS is a validated tool designed to systematically evaluate the severity and intensity of suicidal ideation and behavior.
12-Lead ECG: Mean change from Baseline to End-of-Treatment in QT interval | From Screening to Day 30 and follow up visit 30 days post last dose
12-Lead ECG: Mean change from Baseline to End-of-Treatment in PR interval | From Screening to Day 30 and follow up visit 30 days post last dose
12-Lead ECG: Mean change from Baseline to End-of-Treatment in QRS interval | From Screening to Day 30 and follow up visit 30 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Russell Chin, Study Director — GRIN Therapeutics, Inc.
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd, Brisbane, Queensland
  - Nucleus Network Pty Ltd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No